CLINICAL TRIAL: NCT03210506
Title: The Changes of Cytokines During Pegylated Interferon α-2a and Nucleoside Analogues Treatment in Patients With Chronic Hepatitis B
Brief Title: The Changes of Cytokines During Antiviral Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTXY016
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B Infection
Keywords: chronic hepatitis B; hepatitis B virus; Cytokines; Pegylated Interferon α-2a; Nucleoside Analogues
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): patients who were untreated ever in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly till 48 weeks.
  Interventions: Drug: Peginterferon Alfa-2a
- control group (No Intervention): patients who were untreated ever in immune-active phase took Nucleoside Analogues for maintenance treatment.

INTERVENTIONS:
Drug: Peginterferon Alfa-2a — patients untreated in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly in experiment group.
  Other Names: Peg-IFN-α
  Arms: experimental group

SUMMARY:
Pegylated interferon α-2a(Peg-IFN-α) not only inhibit viral replication, but also play an important role in immune regulation, while Nucleoside analog(ue) drugs only inhibit viral replication. In hepatitis B infection, cytokines played a vital role. This study was aimed at investigating the changes of cytokines during Peg-IFN-αand nucleoside analog(ue) therapy.Meanwhile, the investigators wanted to verify whether Peg-IFN-α therapy resulted in the secretion of cytokines.

DETAILED DESCRIPTION:
Pegylated interferon α-2a(Peg-IFN-α)and Nucleoside analog(ue) drugs can inhibit viral replication , but Peg-IFN-α also play an important role in immune regulation . In hepatitis B infection, cytokines including Fit-3L, IFN-alpha2, IFN-gama, IL-10, IL-17A,IL-2, IL-6, TNF-alpha, TGF-beta1, TGF-beta2,TGF-beta3, played a vital role.Peg-IFN-α recommended as the first-line treatment has a higher chance to achieve HBeAg seroconversion and even HBsAg disappearance than nucleoside analog(ue) drugs, which might be related to the increase of cytokine secretion in the case of hepatitis and during Peg-IFN-α therapy.This study was aimed at investigating the changes of cytokines during Peg-IFN-αand nucleoside analog(ue) therapy.Meanwhile, the investigators wanted to clarify whether Peg-IFN-α therapy led to the secretion of cytokines.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg and HBeAg positive for more than 6 months, HBV DNA detectable with ALT level abnormal lasted for three months and at least time190 IU/L or liver puncture biopsy demonstrated apparent inflammation, never treated before enrolled.

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the changes of cytokines | after treatment 24 weeks
  the changes of cytokines levels will be measured by Luminex test after Pegylated Interferon α-2a and entecavir((ETV) Treatment 24 weeks.

SECONDARY OUTCOMES:
the change of HBVDNA levels (IU/ML) | afte treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBV DNA levels
the change of ALT levels(U/L) | afte treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by ALT levels
the change of AST levels(U/L) | afte treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by AST levels
the change of HBsAg levels (IU/ML) | afte treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBsAg levels
the change of HBeAg levels (IU/ML) | afte treatment 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBeAg levels

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China